CLINICAL TRIAL: NCT00913094
Title: Bioimpedance Evaluation of Therapeutic Titration in Essential, Refractory Hypertension (BETTER-HTN)
Brief Title: Bioimpedance Evaluation of Therapeutic Titration in Essential, Refractory Hypertension
Acronym: BETTER-HTN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: CardioDynamics (Industry)
Responsible Party: Rhonda Rhyne, President, CardioDynamics
Other Study IDs: 07001-M2-1-2-3
Record Dates: First submitted 2009-06-01; First posted 2009-06-03 (Estimated); Last update posted 2009-06-11 (Estimated); Status verified 2009-06

CONDITIONS: Hypertension
Keywords: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- ICG: Group will have results blinded during observational phase of study. Results will be revealed at time of testing during the validation phase of the study.

SUMMARY:
To determine whether impedance cardiography (ICG) parameters can predict favorable or unfavorable blood pressure (BP) response and time to BP control prior to initiation or intensification of specific antihypertensive drug classes and drug combinations, independent of initial BP levels.

DETAILED DESCRIPTION:
* Patients with higher vascular resistance index and/or lower arterial compliance index will lower BP faster and to a greater degree overall when receiving vasodilating agents - such as ACEI's, ARB's, dihydropyridine CCB's, direct vasodilators, and central alpha agonists.
* Patients with an elevated cardiac index will lower BP faster and to a greater degree overall when receiving agents that reduce contractility, heart rate, or blood volume - such as beta blockers, non-dihydropyridine CCB's, and other agents that are known to reduce cardiac index.
* Patients with an elevated thoracic fluid content or lower orthostatic change in thoracic fluid content will lower BP faster and to a greater degree overall when receiving diuretics (thiazide, loop, potassium sparing), however - one of these agents will emerge as a superior alternative to reduce BP in patients with high thoracic fluid content / low orthostatic change in thoracic fluid content.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years of age
* Able to provide written consent
* Meet JNC definition of hypertension
* Lab results with 6 months for: serum creatinine, urine albumin/creatinine ratio, and at least one of the following: serum glucose, or glycated hemoglobin, or hemoglobin A1C

Exclusion Criteria:

* Active cardiovascular disease (unstable angina, stage C or D heart failure, uncontrolled superventricular arrhythmia, hx of ventricular arrhythmia, stroke or TIA within 6 months, ACS within 6 months)
* Implantation of activated ventricular pacemaker
* Known hypersensitivity or allergy to sensor gel or adhesives
* Skin lesions prohibiting sensor placement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited form a population of subjects presenting to a specialty hypertension clinic
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2009-01; Primary Completion 2011-01 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
To determine if ICG can predict therapeutic response to antihypertensive medications | 2009-2010
To confirm derivation phase of ICG prediction to therapeutic response of antihypertensive medications. | 2010-2011

CONTACTS AND LOCATIONS:
Overall Officials: John M Flack, MD, Principal Investigator — Wayne State University, and Detroit Medical Center
Locations (1):
- Wayne State University, Detroit, Michigan, United States